CLINICAL TRIAL: NCT03985280
Title: Randomized Clinical Trial to Evaluate the Efficacy of Two Techniques Against Hip Pain: Cooled Radiofrequency , Compared to Intraarticular Injection.
Brief Title: Radiofrequency Versus Intraarticular Local Anesthestic and Steroids Injection for Chronic Hip Pain.
Acronym: HIPAIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jorge Orduña-Valls (Other)
Responsible Party: Sponsor-Investigator, Jorge Orduña-Valls, Pain physician in Hospital Clínico Universitario de Valencia, Hospital Clínico Universitario de Valencia
Organization: Hospital Clínico Universitario de Valencia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIPAIN
Record Dates: First submitted 2019-02-25; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Hip Pain Chronic
Keywords: Cooled radiofrequency; Radiofrequency; Hip pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cooled radiofrequency (Experimental): The procedure will be performed under regimen of major ambulatory surgery, it will be done under guidance of combined X-ray and ultrasound. . The nerves will be located b, after applying AL (Lidocaine 1%), a RF needle will be placed in the objective position.After verifying the positive sensitive and negative motor responses the cooled radiofrequency will proceed (previous application of local anesthesia (lidocaine 2%)). Cooled RF will be performed for 2:30 minutes at 60 degrees.
  Interventions: Device: Cooled radiofrequency
- Intraarticular local anesthetic and steroids injections (Active Comparator): An intraarticular injection will be done in ambulatory surgery regimen with a 22 Gauge needle. Intraarticular injection will be done under Fluoroscopic guidance (X-rays) with intra articular position confirmation by infusion of iodine contrast (Omnipaque 240). Once the needle position has been verified we will administer 10 mg of bipuvacaine, and 40 mg triamcinolone hexacetonide.
  Interventions: Drug: Intraaticular steroids and local anesthetic injections

INTERVENTIONS:
Device: Cooled radiofrequency — Under guidance of combined X-ray and ultrasound the nerves will be located . After local anesthetic aplication cooled RF needle will be apply in the objective position. Cooled RF will be performed for 2:30 minutes at 60 º C degrees.
  Arms: Cooled radiofrequency
Drug: Intraaticular steroids and local anesthetic injections — Intraaticular steroids and local anesthetic injections
  Arms: Intraarticular local anesthetic and steroids injections

SUMMARY:
Pilot, prospective, randomized study to compare the effectiveness of two techniques against chronic hip pain :cooled radiofrequency on sensory innervation of the hip and intra-articular infiltration of local anesthetic and corticoid.

EudraCT protocol code. 2018-000269-36

Promoter / Principal Investigator. Jorge Orduña Valls

Name of the person responsible for the monitoring:

Nativity Well of the Rose.

Design. Pilot, prospective, randomized study to compare the effectiveness of two techniques against chronic pain of hip: radiofrequency cooled on sensory innervation of the hip and intra-articular infiltration of local anesthetic and corticoid.

Phase of the trial. Phase IV, efficacy evaluation with respect to standard treatment.

Conditions to study. Percentage of subjects with VAS reduction greater than 50% compared to baseline at three months after application of the technique in the two treatment groups.

Longer duration of the analgesic effect (defined as a reduction of the VAS greater than 50% basal) at six months from the application of the technique in patients with hip pain.

Intervention. Application of radiofrequency cooled on nerve endings of the hip. The standard treatment Non-surgical consists of intra-articular injection of local anesthetic and corticoid.

Main and secondary objective.

Main goal:

* Percentage of subjects with improvement in the two groups defined as VAS reduction greater than 50% with respect to the baseline after three months from the application of the technique.
* Compare the persistence of the clinical effect in terms of pain reduction (quantified by a reduction of 50% in the VAS scale compared to the baseline) after six months after the application of the Radiofrequency cooled on sensitive nerve branches of the hip compared to intra-articular injection of local anesthetic and corticoid.

Secondary objectives:

* Compare the improvement of functional capacity of patients submitted to radiofrequency cooled compared to those treated by intra-articular injection of local anesthetic and corticosteroid measured by the WOMAC and Oxford Hip score scales.
* Compare the duration of the clinical improvement in terms of pain reduction quantified by the scale VAS (analog visual scale) per year after the application of both techniques.
* To compare the improvement of the quality of life of patients subjected to radiofrequency cooled with respect to those treated by intra-articular injection of local anesthetic and corticosteroid measured by the SF 36 scale.

Main valuation variable.

Main variable:

The evaluation of pain by means of the Visual analogic scale (VAS) A significant reduction in pain will be considered when VAS decreases by> 50% of the baseline value.

Secondary variables:

* Functional improvement valued by the scales: Oxford Hip score, WOMAC
* Better of the quality of life valued by the SF 36 scale
* The duration of the clinical effect by means of the duration of improvement of the VAS scale.

Population under study and total number of patients. Adult patients with chronic hip pain greater than three months who has not responded to treatment conservative and that is not subsidiary of surgery either by the evolutionary stage or by contraindications related to morbidity terms.

Period of follow-up. The duration of the intervention is 12 months from randomization. After the scheduled interventions, patients will be scheduled for monthly follow-up, three, six and twelve months after the procedure

DETAILED DESCRIPTION:
Pilot, prospective, randomized study to compare the effectiveness of two techniques against chronic hip pain :cooled radiofrequency on sensory innervation of the hip and intra-articular infiltration of local anesthetic and corticoid.

Phase of the trial. Phase IV, efficacy evaluation with respect to standard treatment.

Conditions to study. Percentage of subjects with VAS reduction greater than 50% compared to baseline at three months after application of the technique in the two treatment groups.

Longer duration of the analgesic effect (defined as a reduction of the VAS greater than 50% basal) at six months from the application of the technique in patients with hip pain.

Intervention. Application of radiofrequency cooled on nerve endings of the hip. The standard treatment Non-surgical consists of intra-articular injection of local anesthetic and corticoid.

Main and secondary objective.

Main goal:

* Percentage of subjects with improvement in the two groups defined as VAS reduction greater than 50% with respect to the baseline after three months from the application of the technique.
* Compare the persistence of the clinical effect in terms of pain reduction (quantified by a reduction of 50% in the VAS scale compared to the baseline) after six months after the application of the Radiofrequency cooled on sensitive nerve branches of the hip compared to intra-articular injection of local anesthetic and corticoid.

Secondary objectives:

* Compare the improvement of functional capacity of patients submitted to radiofrequency cooled compared to those treated by intra-articular injection of local anesthetic and corticosteroid measured by the WOMAC and Oxford Hip score scales.
* Compare the duration of the clinical improvement in terms of pain reduction quantified by the scale VAS (analog visual scale) per year after the application of both techniques.
* To compare the improvement of the quality of life of patients subjected to radiofrequency cooled with respect to those treated by intra-articular injection of local anesthetic and corticosteroid measured by the SF 36 scale.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Chronic hip pain (more than 3 months) that has not responded to conservative treatment, therapy pharmacological, physiotherapy or TENS).
* Mechanical pain in the affected limb with a VAS of at least 50 mm during the ambulation
* Patients for whom it is possible to carry out all the scheduled visits of the study, with capacity for go in the established deadlines to the control visits.
* Greater than 50% improvement in the VAS scale after the two anesthetic blocks made with anesthetics local of different duration (bupivacaine 0.25% and mepivacaine 2%)
* Moderate to severe osteoarthrosis determined with grades Kellgren-Lawrence II, III, IV.
* Stable doses of analgesics for at least 30 days before starting the study.
* Patients who have performed the Oxford Hip Score and WOMAC test 3 months or less before the study.
* Absence of allergy or adverse events known to any of the medications administered:

local anesthetics of amide group and iodinated contrasts.

-Negative pregnancy test (women of childbearing age) and commitment to guarantee contraception during the study

Exclusion Criteria:

* Signs of alarm or infection in the joint affects.
* Signs of active infection, immunosuppression or active HIV.
* Severe psychiatric diseases.
* Patient with hip prosthesis.
* Pain added to an unexplained weight loss of more than 5% 90 days or less before the beginning of the study.
* Pain of root origin established in the affected limb, or neurodegenerative diseases of the Peripheral nervous system.
* Patients with basic tumor pathology or who have had cancer in the five years prior to the inclusion.
* Alterations of the coagulation or taking of anticoagulants / antiaggregants (except aspirin 150 or 300) mg / day) at the beginning of the study, which can not be suspended for basic pathology during an interval prudent for the realization of the technique.
* Patient that has participated in a clinical study the previous 30 days in which they are performed interventions that may affect the results of the study.
* Patient with a diagnosis of disorder due to substance abuse or alcoholism.
* Patient who is in process for the award of a disability or degree of disability.
* Pregnant or lactating patient.
* Patient under treatment with opioids with doses greater than the equivalent to 90 milligrams of oral morphine / day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
- Percentage of subjects with improvement measured by VAS after three months. -Compare the persistence of the clinical effect in terms of pain reduction (quantified by a reduction of 50% in the VAS scale compared to the baseline) after six months | 3 months
  VAS --- 100 the most , 0 the less

SECONDARY OUTCOMES:
-Compare the improvement of functional capacity measured by the WOMAC. | 12 months
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68
-Compare the duration of the clinical improvement in terms of pain reduction quantified by the scale VAS (analog visual scale) per year after the application of both techniques. | 12 months
  VAS (analog visual scale)-- 0 the worst, 100 the best
- To compare the improvement of the quality of life of patients subjected to radiofrequency cooled with respect to those treated by intra-articular injection of local anesthetic and corticosteroid measured by the SF 36 scale. | 12 months
  SF 36 scale. 1 the best, 5 the worst
-Compare the improvement of functional capacity measured by the Oxford Hip score . | 12 months.
  12 questions--- 40-48 pints --May indicate satisfactory joint function. May not require any formal treatment.
  Score 0 to 19--May indicate severe hip arthritis. It is highly likely that you may well require some form of surgical intervention, contact your family physician for a consult with an Orthopaedic Surgeon.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital clinico universitario de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No